CLINICAL TRIAL: NCT05112887
Title: Osteopathic Manipulative Therapy Effects on Prolonged Post-COVID Olfactory Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: American Osteopathic Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-F-13
Record Dates: First submitted 2021-11-05; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-03

CONDITIONS: COVID-19 Lower Respiratory Infection; SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Participants will have to email a positive COVID-19 test result >14 days prior to MS861918@ohio.edu. There will be a correspondence with the participant to ask them if they feel their sense is still decreased or absent and then candidacy for study will be determined. 20 participants will be divided randomly into sham OMT treatment groups and real OMT treatments. 10 in each group. Participants will rate on a scale of 0-10 (0 being no smell, and 10 being pre-COVID19 exposure smell) the ability to smell 4 items blindfolded pre-treatment as well as attempt to identify the substance
Who Masked: Participant, Outcomes Assessor
Masking Description: Individual testing smell function was masked to whether participant was in treatment group or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMT Group (Experimental): The OMT protocol treatment sequence was performed in the following order:
  1. Rib raising from a seated position 2. Suboccipital Release from a supine position 3. Thoracic Inlet Release 4. Miller Lymphatic Pump 5. Pedal Pump 6. Suboccipital Release 7. Cranial Sinus Effleurage
  1. Engaging the sagittal midline of occiput with pressure until release of the tissue is palpated
  2. Direct pressure along the external region of the transverse sinus until release of the tissue is palpated.
  3. Pressure on sagittal suture with transverse traction until release of the tissue is palpated
  4. Pressure on metopic suture with transverse traction in a pulsatile manner
  5. Vault hold
  1. Appreciate cranial respiratory motion 2. Diagnose cranial strain pattern 3. Place cranial strain pattern into position of ease
  Interventions: Other: Osteopathic Manipulative Therapy
- Placebo/Light Touch/Sham Group (Placebo Comparator): Participants in the sham/placebo group were lightly touched in equivalent positions to the OMT treatments. First, sham participants were lightly touched on the thoracic cage while seated, followed by light touch of the neck, chest, feet, and cranium while supine. The length of light touch was modeled after the approximate time needed for the OMT matching each treatment region. Each treatment sequence lasted about 20 minutes in total.
  Interventions: Other: Osteopathic Manipulative Therapy

INTERVENTIONS:
Other: Osteopathic Manipulative Therapy — Osteopathic Manipulative Therapy is a type of hands-on manipulative medicine where the physician uses their hands and knowledge of anatomy to encourage the human body to reattain homeostasis.
  Other Names: Osteopathic Manipulative Medicine

SUMMARY:
The goal of this project is to determine the efficacy of a treatment method that increase a participants sense of smell after suffering from COVID-19 related decline in smell. Participants have to be greater than 14 days from positive COVID-19 test and still have a decreased sense of smell. https://jaoa.org/article.aspx?articleid=2765119 this article is a review of literature regarding why OMT can have a positive effect on individuals suffering from COVID-19

Anosmia: Complete loss of smell Hyposmia: Decrease in smell

DETAILED DESCRIPTION:
The goal of this project will be to determine if OMT can return the sense of smell to participants who previously contracted COVID-19.

Participants will have to email a positive COVID-19 test result >14 days prior to MS861918@ohio.edu. There will be a correspondence with the participant to ask them if they feel their sense is still decreased or absent and then candidacy for study will be determined.

20 participants will be divided randomly into sham OMT treatment groups and real OMT treatments. 10 in each group

Participants will rate on a scale of 0-10 (0 being no smell, and 10 being pre-COVID19 exposure smell) the ability to smell the following items blindfolded pre-treatment as well as attempt to identify the substance:

These will be performed with

1. Perfume
2. Red Onion (sliced)
3. Bourbon
4. Orange

Participants in the sham treatment group will receive a non-osteopathic approach to treatment, which will consist of general palpation of head/neck/shoulder region. Participants in the Osteopathic Manipulation Therapy (OMT) group will receive:

* Rib raising
* Suboccipital Release
* Thoracic Inlet Release
* Miller Thoracic Pump
* Pedal Pump
* Cranial OMT, Performed Indirect Vault hold at conclusion

Stevan Walkowski, D.O. will be providing treatment to both the OMT and Sham group.

Participants will rate on a scale of 0-10 (0 being no smell, and 10 being pre-COVID19 exposure smell) to smell the following items blindfolded pre-treatment as well as attempt to identify the substance 10 min post-treatment:

1. Perfume
2. Red Onion (sliced)
3. Bourbon
4. Orange

Participants will be debriefed following the research procedure. They will be informed of potential side effects that is listed in the risks or discomfort category and will be encouraged to drink water following treatment.

Side effects from sham treatment group: Frustration of not re-acquiring sense of smell

Side effects from OMT treatment group: Headache, dizziness, increase secretion (diarrhea, diuresis) from increase in fluid flow, frustration of not re-acquiring sense of smell

Participants in both groups will be told of the side effects of the OMT treatment group and will be encouraged to drink water following treatment.

Benefits from sham treatment group: none

Benefits from OMT treatment group: May have an increase sense of smell post-treatment

Multiple post-COVID19 individuals who lost sense of smell continue to have a decrease sense of smell after surviving the illness. These people have a decreased ability to smell food, drinks and enjoy shared human experiences which can lead to isolation. Individuals who have a decrease sense of smell are also in increased danger due to not being able to smell hazardous events around them i.e. smoke from a fire, gas filling their house from a leaking gas stove, spoiled food etc..

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Positive COVID test greater than 14 days prior
* Self-identify a decrease in smell after the resolution of their infection

Exclusion Criteria:

* Complete smell recovery after resolution of infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Smell Intensity | 10 minutes will elapse between treatment and post-treatment smell testing.
  Participants will smell the 4 substances blindfolded and will rank each one from 0-10, 0 being no smell and 10 be pre-COVID smell. Participant will then be treated either with OMT or placebo and then asked to resmell the same 4 smell substances and rank them on the same scale.
Smell Identification | 10 minutes will elapse between treatment and post-treatment smell testing.
  Participants will smell the 4 substances blindfolded and attempt to identify the smells. Participants will then receive treatment either OMT or Placebo and will smell the same 4 substances while attempting to identify them again. Correct answers were given a score of "1" and incorrect answers were given a smell of "0"

OTHER OUTCOMES:
Quantitative smell experience | 10 minutes will elapse between treatment and post-treatment smell testing.
  Participants were interviewed prior to pre-treatment smell testing to gain a further understanding of how this ailment affects participants on an individual level.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Walkowski, DO, Study Director — Ohio University
Locations (1):
- Ohio University Heritage College of Medicine - Dublin, Dublin, Ohio, United States